CLINICAL TRIAL: NCT07212751
Title: Coronary CT Angiogram - Prognostic Value of Adverse Plaque Features in Guiding Treatment (CT-PLAQUE)
Acronym: CT-PLAQUE
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW20-057
Record Dates: First submitted 2025-07-07; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-06

CONDITIONS: Determining if the Presence of Adverse Plaque Features Identified From the CT Angiogram Can Help Determining Prognosis and Guide Treatment Options
Keywords: CTCA; CT; Coronary CT; Calcium Score; Plaque; Coronary Artery Disease; CAD; Chest pain; Patients with suspicion of coronary artery disease
MeSH Terms: conditions — Plaque, Amyloid; Coronary Artery Disease; Chest Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient who is ≥ 18 years old presented with chest pain and has undergone CTA before treatment
  Interventions: Diagnostic Test: CTCA

INTERVENTIONS:
Diagnostic Test: CTCA — Patient who is ≥ 18 years old presented with chest pain and has undergone CTA between 01-Jan-2012 and 31-Dec-2022 before treatment
  - If multiple CTAs are taken, the most updated one before treatment commencement will be chosen.

SUMMARY:
The study aims at determining if the presence of adverse plaque features identified from the CT angiogram can help determine prognosis and guide treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is ≥ 18 years old presented with chest pain and has undergone CTA between 01-Jan-2012 and 31-Dec-2022 before treatment
* If multiple CTAs are taken, the most updated one before treatment commencement will be chosen.

Exclusion Criteria:

* Patient who did not undergo cardiac CT scan due to inability to undergo cardiac CT scanning, kidney failure (serum creatinine >250 μmol/L or estimated glomerular filtration rate <30 mL/min), major allergy to contrast.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 28000
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death and all-cause death | 5 years after CTCA examinations

SECONDARY OUTCOMES:
Total plaque, total calcified plaque, total non-calcified plaque, CT-FFR | 5 years after CTCA examinations

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong